CLINICAL TRIAL: NCT01993602
Title: COMPARISON OF LUNG EXPANSION TECHNICS ON THORACOABDOMINAL MECHANICS AND THEIR INFLUENCE ON THE INCIDENCE OF PULMONARY COMPLICATIONS AFTER ABDOMINAL SURGERY: A RANDOMIZED AND CONTROLLED CLINICAL TRIAL
Brief Title: Lung Expansion Technics on Chest Wall Mechanics and Preventing Pulmonary Complication After Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0150/11; FAPESP (Other Grant/Funding Number: 2010/50120-4)
Record Dates: First submitted 2013-11-08; First posted 2013-11-25 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2013-11

CONDITIONS: Surgical Procedure, Unspecified
Keywords: general surgery; postoperative care; breathing exercises; respiratory muscle; postoperative complications; lung volume measurements; pulmonary ventilations; thoracic wall
MeSH Terms: conditions — Postoperative Complications | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Control group (No Intervention): no intervention was performed in this group during postoperative period,
- volumetric incentive spirometry (Active Comparator): patients performed breathing exercises using volumetric incentive spirometer during five postoperative days
  Interventions: Procedure: Breathing exercises
- Flow oriented incentive spirometry (Active Comparator): patients performed breathing exercises using flow oriented incentive spirometer during five postoperative days
  Interventions: Procedure: Breathing exercises
- Deep breathing group (Active Comparator): patients performed deep breathing exercises without any device during five postoperative days
  Interventions: Procedure: Breathing exercises
- Continuous positive airway pressure group (Active Comparator): patients performed breathing exercises using continuous positive airway pressure group during five postoperative days
  Interventions: Procedure: Breathing exercises

INTERVENTIONS:
Procedure: Breathing exercises — The intervention groups (CPAP, VIS, FIS and DB) used the specific device (or not) according to the group allocation.
  The intervention was performed 3 times per day, from 1 to 5 postoperative day. Patients performed 5 sets of 10 repetitions of the specific breathing exercise, with 30 seconds rest between each set.
  The sessions were held in the morning, early afternoon and early evening, always supervised by a physiotherapist.
  Before starting each session, the patient reported the sensation of pain, and if he quantify pain intensity more than 3 in the visual numeric scale (0 to 10) was asked the doctor to administer analgesics aiming that him to perform properly the breathing exercise.
  Arms: Continuous positive airway pressure group; Deep breathing group; Flow oriented incentive spirometry; volumetric incentive spirometry

SUMMARY:
The lung expansion techniques are widely used to prevent postoperative pulmonary complications. However, the effect of each technique on thoracoabdominal mechanics after abdominal surgery and if it influences the rate of postoperative pulmonary complications remains unknown. The investigators hypothesis is that the lung expansion technique that more increases lung volume after abdominal surgery, will be the most efficient in preventing postoperative pulmonary complication after abdominal surgery. The investigators objectives will be to compare the effect of different lung expansion techniques on lung volumes and activation of inspiratory muscle, and prevention of pulmonary complications in patients undergoing upper abdominal surgery. This study will involve 171 patients undergoing elective abdominal surgery. Patients will be randomly divided into 5 groups: no therapy group (n=35), continuous positive airway pressure (CPAP, n=34); volumetric incentive spirometry (VIS, n=34); flow oriented incentive spirometry (FIS, n=33) and deep breathing (DB, n=35). The thoracoabdominal mechanics will be assessed before and 3 days after surgery. Complications will be evaluated by a researcher who did not know to which group each patient belongs.

DETAILED DESCRIPTION:
The assessments performed were thoracoabdominal kinematics (by optoelectronic pletysmography)and respiratory muscles activity (by surface electromyography). The follow pulmonary complications were considered: pneumonia, tracheobronchitis, atelectasis and acute respiratory failed

ELIGIBILITY:
Inclusion Criteria:

* candidates for elective upper abdominal surgery expected to last longer than 120 minutes
* absent of spine or thoracic deformity
* no previous lung parenchyma resection
* no tracheostomy
* able to understand and perform the maneuvers proposed.

Exclusion Criteria:

* cancellation of surgery
* mechanical ventilation for more than 24 hours in the postoperative period
* need for chest tube use
* postoperative cardiac complications
* surgical complication
* reoperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2011-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
thoracoabdominal volume | third postoperative day
  thoracoabdominal volume was evaluated by kinematics (optoelectronic plethysmograph)

SECONDARY OUTCOMES:
postoperative pulmonary complication | participants will be followed for the duration of hospital stay, an expected average of 10 days
  evaluation of pulmonary complications was performed according to pre-established criteria in the research project

OTHER OUTCOMES:
activity inspiratory muscles | third postoperative day
  evaluation was performed by surface electromyography

CONTACTS AND LOCATIONS:
Overall Officials: Celso R Carvalho, PhD, Principal Investigator — School of Medicine of University of Sao Paulo
Locations (1):
- Hospital of Clinics of School of Medicine of University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Lunardi AC, Paisani DM, Silva CCBMD, Cano DP, Tanaka C, Carvalho CRF. Comparison of lung expansion techniques on thoracoabdominal mechanics and incidence of pulmonary complications after upper abdominal surgery: a randomized and controlled trial. Chest. 2015 Oct;148(4):1003-1010. doi: 10.1378/chest.14-2696. PMID 25973670